CLINICAL TRIAL: NCT05093959
Title: Metformin for Older Patients With Heart Failure With Preserved Ejection Fraction
Acronym: Met-PEF
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: University of South Florida (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00076663; U01AG076928 (NIH)
Record Dates: First submitted 2021-10-22; First posted 2021-10-26 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure With Preserved Ejection Fraction
Keywords: heart failure, metformin, inflammation
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, investigators, and outcomes assessors will be unmasked at the end of data collection of all participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin (Active Comparator): 20 weeks of metformin 1500 mg daily. Metformin is a widely used medication with an excellent safety profile. Dosing will be escalated during the first 3 weeks of treatment. Dosing will be initiated with 500 mg taken orally once daily in the evening for 1 week. After one week, the participant will be called to assess tolerance and will be asked to increase dose to two capsules per day for a total 1000 mg per day for one week. At the end of the second week, participants will be called again and if they tolerated the increased dose will be instructed to increase to three capsules (1500 mg/day) per day for the remainder of the 20 weeks. An extended release formulation will be used which improves compliance and reduces GI side effects.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): 20 weeks of placebo 1500 mg daily. Placebo is a biologically inert substance placed in capsules to match appearance of active intervention (metformin). Dosing will be escalated during the first 3 weeks of treatment. Dosing will be initiated with 500 mg taken orally once daily in the evening for 1 week. After one week, the participant will be called to assess tolerance and will be asked to increase dose to two capsules per day for a total 1000 mg per day for one week. At the end of the second week, participants will be called again and if they tolerated the increased dose will be instructed to increase to three capsules (1500 mg/day) per day for the remainder of the 20 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — An extended release formulation will be used which improves compliance and reduces GI side effects.
  Other Names: metformin XR
  Arms: Metformin
Drug: Placebo — Placebo is a biologically inert substance placed in capsules to match appearance of active intervention
  Arms: Placebo

SUMMARY:
Met-PEF will be a randomized, double-blind, placebo-controlled trial to examine the effects of 20 weeks of 1500 mg/day of metformin on physical function, quality of life (QOL), microbiome diversity, leaky gut, and systemic inflammation in patients with 86 older patients with heart failure with preserved ejection fraction (HFpEF).

DETAILED DESCRIPTION:
Enrollment of participants will be conducted at both Wake Forest and Atrium Health (approximately 43 participants at each site) following assessment of eligibility criteria and willingness to participate in the trial. Eligibility criteria are designed to target the population under study and exclude participants unable to safely take the study intervention or undergo study procedures. Informed consent will be obtained from qualified participants. Participants will complete baseline assessments before masked, random assignment to metformin or placebo. The assigned study medications will be dispensed by the research pharmacy. Participants will take assigned metformin or placebo for a treatment period of 20 weeks, starting at 500mg/day and escalating over the first 3 weeks to a target dose of 1500mg/day. Participants will be contacted every 2 weeks for assessment of adverse events, side effects, and adherence. At week 4, participants will be seen in clinic for safety laboratory assessments. At week 20, participants will complete follow-up assessments by an assessor blinded to treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure with preserved ejection fraction (HFpEF) will be defined in accord with the American College of Cardiology/American Heart Association 2013 guidelines statement on Management of heart failure and as previously described. The 4 key inclusion criteria for HFpEF include: 1) clinical signs and symptoms as scored by National Health and Nutrition Examination Survey (NHANES)-HF Clinical Score ≥3 and the Rich Criteria; 2) a normal left ventricular (LV) ejection fraction (≥50%) by echocardiography; 3) LV diastolic dysfunction > grade 1 (American Society of Echocardiography Recommendations); 4) no evidence of significant ischemic, valvular, pulmonary or other medical disorder to account for their symptoms.
* Age ≥60
* Stable HF symptoms and medications for ≥3 weeks
* Final eligibility will be based upon all information available at the conclusion of the baseline visits tests, including review of hospital and outpatient records, history, physical examination, echocardiogram, and familiarization/screening exercise test by a board-certified investigator cardiologist who have extensive experience in heart failure investigations in older persons with HFpEF

Exclusion Criteria:

* History of treatment with metformin or other anti-diabetic drug intended to treat diabetes
* Body mass index (BMI) <25.0
* Uncontrolled dysrhythmia
* Uncontrolled hypertension (systolic blood pressure [SPB]>200 mmHg or diastolic blood pressure [DBP]>100 mmHg at rest)
* Significant anemia (<9.5 g hemoglobin [Hb]) (eligibility will be determined by complete blood count)
* Significant renal insufficiency (estimated glomerular filtration rate [eGFR] <45 ml/min/1.73 m2) (eligibility will be determined by comprehensive metabolic panel)
* Acute or chronic metabolic acidosis
* Type 2 diabetes, or HbA1c>6.5
* Low vitamin B12 (<232 pg/mL)
* Known valvular heart disease, infiltrative cardiomyopathy, or hypertrophic obstructive cardiomyopathy with active obstruction as the primary etiology of HF
* Evidence of significant chronic obstructive pulmonary disease (COPD) defined as either: a. On continuous home oxygen therapy for COPD; b. Hospitalization for COPD in last 6 months
* Any condition that in the judgement of the investigator precludes participation in study or study procedures such as significant dementia, mobility impairment, uncontrolled psychiatric disease, etc.
* Alcohol abuse (>14 drinks/week)
* Current or recent cancer, or chemotherapy/radiation treatment
* Pregnancy-women of child-bearing potential are excluded from participation in this study.
* A treadmill exercise test revealing: a. Evidence of significant ischemia; b. Electrocardiogram: 1mm flat ST depression; c. Stopped exercising due to chest or leg claudication or any reason other than exhaustion/fatigue/dyspnea; d. Exercise SBP > 240 mmHg, DBP > 110 mmHg ; e. Unstable hemodynamics or rhythm; f. Unwilling or unable to complete adequate exercise test
* Exclusions for microbiome testing: a. Antibiotics use within last 30 days; b. Diarrhea and/or vomiting within last 30 days; c. Surgery related to gut in last 6 months; d. Inflammatory bowel disease (such as Crohn's disease or ulcerative colitis), or irritable bowel syndrome
* Plans to leave area within 1 year
* Currently participating in other investigational study
* Refuses informed consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-12-18 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Peak VO2 | Week 20
  Peak VO2 (ml of O2 relative to kg of body weight per minute [ml/kg/min]) is a measure of peak oxygen capacity during exercise, is a standardized, objective, reproducible and valid measure of exercise capacity.

OTHER OUTCOMES:
C-reactive protein | Week 20
  Inflammatory marker in serum blood
Interleukin-6 | Week 20
  Inflammatory marker in serum blood
Tumor necrosis factor-alpha | Week 20
  Inflammatory marker in serum blood
Kansas City Cardiomyopathy (KCCQ) Overall Score | Week 20
  The KCCQ overall score is the main summary score of the KCCQ containing physical, symptom, quality of life, and social subdomains. It is measured on a scale of 0-100 units with higher score indicating better HF-disease-specific quality of life.
Short Physical Performance Battery (SPPB) | Week 20
  The SPPB is a valid, clinically meaningful measure of physical function in older adults. The SPPB has 3 components: standing balance, 4-meter walk, and repeated chair rises, corresponding to balance, mobility, and functional strength. Each component is scored on a scale of 0-4 for a total score of 0-12 units with a higher score indicating better physical function.
6-minute walk distance (6MWD) | Week 20
  6MWD is the distance walked in 6 minutes, with higher distance indicating better function. The 6MWD test is a well-established outcome measure in heart failure. It is valid and reproducible in patients with a wide range of physical function, predicts clinical events, and responds to interventions.
Lipopolysaccharide binding protein (LBP) | Week 20
  LBP is a marker of microbial translocation, is increased in older persons and is related to their reduced physical function.
Fecal Mucin | Week 20
  Fecal mucin (mg/g) is a protein that indicates the mucus barrier functions and mucin production, measured by ELISA assays in feces. The higher the fecal mucin, better the mucus barriers are, or vice-versa.

CONTACTS AND LOCATIONS:
Overall Officials: Dalane W. Kitzman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Atrium Health Sanger Heart and Vascular Clinic Institute, Charlotte, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No
No data are to be shared from this study.